CLINICAL TRIAL: NCT01374750
Title: A Randomized Phase Ⅱ, Trial With Sirolimus-containing Versus mTOR-inhibitor Free Immunosuppression in Patients Undergoing Living Donor Liver Transplantation for Hepatocellular Carcinoma Exceeding Milan Criteria
Brief Title: Efficacy of Sirolimus In Liver Transplantation for Hepatocellular Carcinoma (HCC)
Acronym: Sirolimus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Kwang-Woong Lee, general surgery professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KWLee1004-052-316; H-1004-052-316 (Registry Identifier: H-1004-052-316)
Record Dates: First submitted 2011-04-21; First posted 2011-06-16 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sirolimus; Tacrolimus; Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- m-TOR inhibitor free (Active Comparator): Immunosuppressive drug
  Interventions: Drug: m-TOR inhibitor free
- Sirolimus (Experimental): Immunosuppressive drug
  Interventions: Drug: Sirolimus

INTERVENTIONS:
Drug: Sirolimus — Sirolimus
  Other Names: Rapamune
  Arms: Sirolimus
Drug: m-TOR inhibitor free — calcineurin inhibitors
  Other Names: Tacrolimus; Cyclosporine
  Arms: m-TOR inhibitor free

SUMMARY:
The purpose of this study is to evaluate the anti-tumor effect of sirolimus-based immunosuppressive regimen in patients following living donor liver transplantation for hepatocellular carcinoma exceeding Milan criteria with respect to recurrence-free survival.

DETAILED DESCRIPTION:
The Milan criteria were adopted in most of western countries for deceased donor allocation because they identify a subgroup of candidates with hepatocellular carcinoma (HCC) for whom transplant results are similar to those in patients transplanted for end- stage liver disease without HCC. There is a debate involving expanding the indications beyond the Milan criteria in living donor liver transplantation (LDLT). Some transplant surgeons argue that despite the poorer results, LDLT for advanced HCC may be justified, since donors voluntarily accept the risks of donor hepatectomy to dedicate a graft for HCC patients, who may otherwise have no effective treatment. Especially, in Korea where living donor liver transplantation (LDLT) is commonly performed, the expansion of Milan criteria is inevitable. Sirolimus is a macrolide antibiotic produced by Streptomyces hygroscopic that has demonstrated potent immunosuppressive activity in a number of studies. The efficacy of sirolimus as immunosuppressives has been demonstrated in randomized clinical trials in kidney transplantation. The use of sirolimus in liver transplantation is rapidly increasing from the standpoint of reducing the conventional calcineurin inhibitor toxicity. Sirolimus emerged as an effective alternative for patients with renal insufficiency related to calcineurin inhibitor toxicity. In recent studies, no differences have been observed with respect to rejection or major complications.The use of sirolimus in transplant patients is associated with a dose-dependent increase in serum cholesterol and triglycerides that may require treatment. In recent studies in liver transplant recipients using sirolimus as part of a primary immunosuppressive regimen, the occurrence of acute cellular rejection is relatively low. There is data suggesting that sirolimus is associated with hepatic artery thrombosis. Numerous current studies have shown that sirolimus may have inhibitory effects on the development of cancer. Immunosuppressive agent with antineoplastic activity is inherently attractive in the setting of liver transplantation for HCC. If sirolimus shows some degree of anti-tumor effect in transplant recipients with advanced HCC, the indication of LDLT for advanced HCC can be expanded.Our hypothesis is that sirolimus based-regimen will improve the HCC recurrence free survival. If sirolimus-based protocol shows better recurrence free survival, the indication of LDLT for HCC can be expanded. LDLT can be one of the best treatment modalities for advanced HCC. The patients with advanced HCC can have benefit by liver transplantation.

ELIGIBILITY:
Inclusion Criteria :

1. Age ≥ 18 yrs and weight ≥ 40 kg.
2. Histologically proven HCC exceeding Milan criteria before randomization, regardless of the prior therapy
3. Signed and dated written informed consent
4. Lack of relevant exclusion criteria
5. Women who were of childbearing potential must have had a negative qualitative serum pregnancy test before Investigational agent administration and must have agreed to use a medically acceptable method of contraception during treatment period of the study.

Exclusion Criteria :

1. Multiple organ recipients
2. Deceased donor liver transplant
3. Known hypersensitivity to Simulect®, sirolimus, tacrolimus, cyclosporine, or MMF or its derivatives
4. Hyperlipidemia refractory to optimal medical management (cholesterol >300 mg/dl; Triglycerides > 350 mg/dl)
5. Evidence of significant local or systemic infection at the time of randomization.
6. Known HIV-positive patients
7. Women of child-bearing potential not willing to take contraception
8. Patients with non-HCC malignancies within the past 5 years, excluding successfully treated squamous cell carcinoma and basal cell carcinoma of the skin
9. Patients with HCC involvement of a major branch(portal vein, hepatic vein, etc.) of any hepatic blood vessel on pathological evaluation c.f. Major branch is defined as the first or the second order branch (e.g. In case of the portal vein, right and left portal vein, right anterior and posterior portal vein, and left medial and lateral portal vein)
10. Patients with any evidence of extrahepatic HCC metastasis
11. Patients with a psychological, familial, sociologic or geographic condition potentially hampering compliance with the study protocol and follow-up schedule
12. Use of any investigational drug or treatment up to 4 weeks before enrolling in the study and during the 24-month treatment period.
13. Hepatic artery stenosis or occlusion diagnosed by Doppler
14. Patients with severe renal insufficiency at randomization time point (GFR < 40mL/min, Proteinuria > 800mg/24hrs)
15. Patients with severe leucopenia and/or thrombocytopenia refractory to medical treatment (ANC < 500/ul,platelet < 30K/ul)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2010-05; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
To evaluate recurrence-free survival | 3 years
  To evaluate the anti-tumor effect of sirolimus-based immunosuppressive regimen in patients following living donor liver transplantation for hepatocellular carcinoma exceeding Milan criteria with respect to recurrence-free survival

SECONDARY OUTCOMES:
To evaluate the survival rate | 3 years
  The recurrence is defined by tumor recurrence in imaging study. The recurrence free survival will be calculated by Kaplan-Meier method.
To evaluate the renal function | 3 years
  Renal function will be evaluated by calculated GFR (Cockcroft-Gault method) at postoperative 6month, 12month, 18month, 24month, 30month, and 36month.
To evaluate the safety with sirolimus | 3 years
  Safety of sirolimus will be evaluated by the comparison of proportion of patients with serious adverse events during the follow-up period between two groups (m-TOR goup vs. m-TOR free group). Other minor side effects will be monitored and compared between two groups as well.

CONTACTS AND LOCATIONS:
Overall Officials: Kwang-woong Lee, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea